CLINICAL TRIAL: NCT06624891
Title: Evaluation of Perioperative Fluid Responsiveness in Neurosurgery: Interest of the Pleth Variability Index
Brief Title: Interest of the Pleth Variability Index in Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurology, Tunisia (Other)
Responsible Party: Principal Investigator, Hammami Rabeb, university hospital assistant, National Institute of Neurology, Tunisia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PVI IN NEUROSURGERY
Record Dates: First submitted 2024-08-22; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-08

CONDITIONS: Intraoperative Monitoring; Hypovolemia; Fluid Challenge
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Intervention Model Description: prospective comparative randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pleth variability index (PVI) (Experimental): Participants will be monitored during the intervention using a Radical-7 Pulse CO-Oximeter to instantly determine the pleth variability index (PVI). If the PVI is more than 14% for at least 5 minutes, 250 ml of gelofusine solution will be given over 10 minutes.
  Interventions: Other: perioperative fluid responsiveness with the Pleth variability index
- delta PP (Active Comparator): Participants will be monitored during the intervention using arterial catheter to instantly determine delta PP. If Delta PP is more than 13% for at least 5 minutes, 250 ml of gelofusine solution will be given over 10 minutes.
  Interventions: Other: perioperative fluid responsiveness with delta PP

INTERVENTIONS:
Other: perioperative fluid responsiveness with the Pleth variability index — Perioperative fluid challenge and responsiveness will be based on monitoring the pleth variability index. In fact, volemia will be estimated with the PVI.
  Arms: pleth variability index (PVI)
Other: perioperative fluid responsiveness with delta PP — fluid challenge and responsiveness during intervention will be based on monitoring delta PP.
  Arms: delta PP

SUMMARY:
This clinical trial aims to study the interest of the Pleth Variability Index (PVI) to evaluate perioperative fluid responsiveness in neurosurgery in adults.

The main question it aims to answer is:

• Does the Pleth variability index predict fluid responsiveness in neurosurgery? Researchers will compare the Pleth variability index to dela PP to see if it predicts fluid responsiveness in neurosurgery.

Once participants give their consent, they will be randomly assigned to one of two groups. In one group, fluid responsiveness will be monitored using the Pleth Variability Index, while in the other group, it will be monitored using delta PP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients proposed for intracranial surgery
2. Must be aged 18 and over
3. Must be classified as ASA I, ASA II, and ASA III according to the American Society of Anesthesiologists classification

Exclusion Criteria:

1. Non-consenting patients
2. Patients classified ASA IV or higher
3. Cardiac arrhythmia
4. Heart disease with left ventricular ejection fraction less than 45%
5. Obesity with a BMI greater than 40 Kg/m2.
6. Peripheral vascular disease
7. Severe lung disease
8. End-stage renal disease
9. Intraoperative cardiac arrhythmia
10. The occurrence of cardiac arrest
11. The occurrence of hemorrhagic shock
12. Intraoperative use of low tidal volumes or high respiratory rates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Value of PVI in fluid responsiveness in neurosurgery | chanfe of PVI value from baseline to a value more than 14% and untill the end of surgery
  Investigate the value of the plethysmographic variability index (PVI) in assessing the response to perioperative vascular filling in neurosurgery.

SECONDARY OUTCOMES:
Amount of fluids administered intraoperatively | during the surgery
Renal, metabolic and hydroelectrolytic repercussions. | up to the first 24 hours postoperatively
Length of postoperative stay | up to hospital discharge, an average of 4 days
Incidence of post-operative complications | up to hospital discharge, an average of 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurologie Mongi Ben-Hamida, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided